CLINICAL TRIAL: NCT00372346
Title: Safety and Efficacy Study of Transplantation of EPCs to Treat Idiopathic Pulmonary Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 419000-X90305
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2006-09-06 (Estimated); Status verified 2006-08

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

INTERVENTIONS:
Procedure: Transplantation of autologous endothelial progenitor cells

SUMMARY:
Experimental data suggest that transplantation of endothelial progenitor cells (EPCs) attenuates monocrotaline-induced pulmonary hypertension in rats and dogs. In addition, clinical studies suggest that autogolous progenitor cells transplantation is feasible and safe in patients with ischemic disease. This study will investigate the feasibility, safety, and initial clinical outcome of intravenous infusion of autologous EPCs in patients with idiopathic pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic pulmonary arterial hypertension

  1. in New York Heart Association (NYHA) functional class II to III
  2. a mean pulmonary artery pressure more than 30 mmHg on right heart catheterization
  3. the ability to walk ≥50 m during a standardized 6-minute walk test

Exclusion Criteria:

* Pulmonary hypertension as a result of heart disease, pulmonary disease, sleep-associated disorders, chronic thromboembolic disease, autoimmune or collagen vascular disease, HIV infection, liver disease, NYHA functional class IV, major bleeding requiring blood transfusion, diabetes, renal dysfunction, and evidence for malignant diseases were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-06; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: junzhu chen, MD, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Cardiology, the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Takahashi M, Nakamura T, Toba T, Kajiwara N, Kato H, Shimizu Y. Transplantation of endothelial progenitor cells into the lung to alleviate pulmonary hypertension in dogs. Tissue Eng. 2004 May-Jun;10(5-6):771-9. doi: 10.1089/1076327041348563. PMID 15265294